CLINICAL TRIAL: NCT00289055
Title: A Clinical Investigation of the SMART™ Nitinol Self-Expandable Stent Versus Balloon Angioplasty for the Treatment of Superficial Femoral Artery Occlusions
Brief Title: The Study to Compare the Treatment of Angioplasty and Stents in SFA Occlusions.
Acronym: DURAVEST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Medical Affairs Director, Cordis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EE04-01NL
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Arterial Occlusive Diseases
Keywords: Peripheral Artery Occlusive Disease
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Arterial Occlusive Disease 1 | interventions — Stents; Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cordis SMART™ Nitinol Stent
  Interventions: Device: stent
- 2 (Active Comparator): balloon angioplasty
  Interventions: Device: angioplasty

INTERVENTIONS:
Device: stent — Cordis SMART™ Nitinol Stent
  Arms: 1
Device: angioplasty — balloon angioplasty
  Arms: 2

SUMMARY:
The main objective of this study is to assess the patency rate of the nitinol self-expandable stent device in the treatment of superficial femoral artery (SFA) occlusions as compared to angioplasty only.

DETAILED DESCRIPTION:
This is a multi-center prospective, randomized, two-arm study evaluating performance of the Cordis SMART™ nitinol self-expanding stent as compared to balloon angioplasty only. Patients will be randomized on a 1:1 basis. It is anticipated that a total of 120 patients will be entered into the study.

The study population will consist of symptomatic peripheral vascular disease patients with SFA occlusions. The disease will consist of symptomatic, long de novo or restenotic occlusions (5 - 14.5 cm) on diagnostic imaging with a history of at least 6 months. The occlusions must not extend beyond the proximal popliteal artery. For the purpose of this protocol, no lesion within 3 cm of the upper part of the patella may be treated. The distal popliteal artery must be patent with no hemodynamic stenosis as well as two calf vessels. Reference vessel diameter must be >= 4.0 to <= 6.0 mm.

Trial participants will be randomized to the SMART™ nitinol self-expanding stent or to balloon angioplasty only.

Patients will be followed for twelve months post-procedure. Study examinations will be done at screening, procedure time, discharge, six, and twelve months post procedure.

This study will be conducted at 8 investigational sites in The Netherlands.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic leg ischemia by Rutherford Classification (category 1, 2, 3, 4 or 5); duration of intermittent claudication (category 1-3) should be at least 6 months
2. The patient should be suitable for percutaneous transluminal angioplasty (PTA) and also for stenting.

Exclusion Criteria:

1. Poor aortoiliac or common femoral "inflow", which would be deemed inadequate to support a femoropopliteal bypass graft.
2. Patient having total occlusions or severe stenosis of the iliac artery on the same side must be excluded.
3. Gangrene in index limb (Rutherford category 6).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Primary patency. | 12 months

SECONDARY OUTCOMES:
Technical success defined as a successful access and deployment of the device with recanalization, determined by angiography. | at deployment
Procedural success defined as successful recanalization, without the occurrence of a SAE. | up to the moment haemostasis has been achieved
Procedural complications, defined as any adverse event | from start of the procedure up to the moment haemostasis has been achieved
Ankle Brachial Index. | discharge and 12 months
Treadmill test. | 12 months
Restenosis measured by Duplex Ultrasound. | 12 months
Quality of Life assessment. | baseline, 6, and 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jim Reekers, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- AMC, Amsterdam, Netherlands